CLINICAL TRIAL: NCT04218643
Title: Ultrasound-guided Peripheral Intravenous Catheter Insertion Technique and the Effects on Overall Site Utilization and Failure
Brief Title: Ultrasound-guided Peripheral Intravenous Catheter Insertion Technique
Acronym: PIVC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too difficult due to lost staff after COVID
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 042-19
Record Dates: First submitted 2019-11-07; First posted 2020-01-06 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2021-11

CONDITIONS: Catheterization, Peripheral Venous; Phlebitis; Infiltration
Keywords: peripheral intravenous catheter; ultrasound-guided; IV insertion; catheter to vein ratio
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: Randomized prospective trial comparing US-guided PIVC insertion with standard PIVC insertion technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard technique (Active Comparator): Intravenous catheter inserted via standard technique
  Interventions: Other: Standard technique
- Ultrasound-guided technique (Experimental): Intravenous catheter inserted via ultrasound guidance
  Interventions: Other: Ultrasound-guided technique

INTERVENTIONS:
Other: Ultrasound-guided technique — IV inserted via ultrasound guidance
  Arms: Ultrasound-guided technique
Other: Standard technique — IV inserted via standard technique
  Arms: Standard technique

SUMMARY:
This comparative treatment study aims to challenge a current clinical practice. Specifically, whether the use of ultrasound-guided peripheral intravenous catheter insertion results in lower post insertion failure rates with longer utility time compared to peripheral intravenous catheters (PIVC) inserted in the standard manner during the emergency department (ED), observation and in-patient stay. There are two secondary aims to the study: a) determining if ultrasound-guided peripheral intravenous catheter insertion results in lower post removal complication rates compared to PIVCs inserted in the standard manner; and b) determining if catheter-to-vein ratio can predict post insertion success of PIVCs and what catheter-to-vein ratio is most successful. In this study, catheter-to-vein ratio is defined as the diameter of the lumen of the vein divided by the outside diameter of the catheter.

DETAILED DESCRIPTION:
This study is a randomized prospective trial comparing US-guided PIVC insertion with standard PIVC insertion technique. This study will evaluate the predictive strength of catheter-to-vein ratio to PIVC post insertion success.

The study population is all patients presenting to the ED. The sample population will be patients requiring a PIVC for treatment or diagnostic purposes and don't have an existing PIVC (EMS or other). Inclusion and exclusion criteria focusing on most suitable participants and safety will determine the participant population. Participants will be randomized to one of two cohorts; 1) PIVC insertion based on standard technique and 2) US-guided PIVC insertion.

There will be two data collection phases in this study:

Phase one occurs in the emergency department (ED). ED staff will be notified of the study period, however to minimize bias, details of the study will not be given. Patients in this phase include those registered in the ED seeking treatment. To identify potential candidates, the investigator will perform an initial screening by communicating with ED staff. Initial screenings will be recorded without using any identifying data. When a potential participant is identified, the investigator will then coordinate with ED staff, approach the candidate and confirm that they meet inclusion and exclusion criteria. If the patient qualifies for enrollment, the investigator will review the study purpose including risks and benefits of enrolling, and have the patient sign the consent form. Randomization will occur after obtaining consent. Patients will have a PIVC inserted by any qualified Nurse or Medic. The PIVC will be placed according to the Reading Hospital Peripheral Intravenous Therapy for Adults guideline. After the PIVC (Standard or US-guided) is inserted, the investigator will then measure the vein prior to any infusion that could distort vein measurement.

All investigators involved with vein measurement will complete vein measurement training. The vein size will be measured using one of the following US machines: SonoSite Edge II or X-Porte each equipped with a 13-6 MHz, 6 cm linear probe (FUJIFILM SonoSite, Inc. Bothell, WA, USA). The investigator will then record collected data on the phase one data collection form and place the form in a secure container. A member of the research team will then collect the completed data collection forms and enter the data in a secured study database. To limit bias, investigators will not inform the ED staff of the specifics of this study and will only provide enough information for data to be collected safely and accurately. In the event that a PIVC could not be successfully inserted according to the randomized technique, the PIVC will be analyzed in an intention to treat (ITT) format and the participant will receive vascular access as per the treatment team.

Phase two of data collection is divided into two parts, and participants in this phase include those that had a PIVC inserted by either randomized method and were subsequently placed in an observation status, inpatient status or discharged home. Phase two part one occurs after the PIVC has been removed. Data collection is performed electronically and may also involve verbal follow up. Trained investigators will obtain an active list of subjects whose PIVC was removed. Each subject will have a blank phase two part one data collection form completed in its entirety when possible. Subjects who remain on an inpatient or observation status will be followed in the electronic health record (EHR). In this study post insertion failure is identified when any of the following reasons for PIVC removal has been entered into the participants EHR: leakage, drainage, phlebitis, painful, occluded, infiltrated, and catheter damage. If more than one of these reasons has been entered, the investigator will further investigate the EHR to determine the primary reason for removal. If electronic data is not sufficient and the subject is still hospitalized, the investigator will attempt to visit the subject for completion of data collection. Completed phase two part one forms will be placed in a secure container until entry into the study database. Following data entry, paper forms involved in this part will be destroyed. Subjects with a PIVC that was removed for a reason not determined as a failure will proceed into phase two part two.

Phase two part two occurs when a PIVC was removed without complication. A trained investigator will obtain a list of subjects whose PIVC was removed without complication. The investigator will determine if 48 hours has passed since the removal of the PIVC. If so, a post removal follow-up interview is performed if the patient is still admitted in the hospital or a phone interview is conducted if the patient was discharged home. Participant charts will also be reviewed for any subsequent ED or primary care physician visits related to PIVC complication(s). The investigator completes the phase two part two data collection form and places it in a secured container. A time limit of 48 hours to contact the participant has been set for this study. A member of the research team will then collect the data collection forms and enter the data in the secured study database.

Statistics and data analysis

Sample size calculation:

The baseline failure rate for post-insertion PIVCs at Reading Hospital is 30%. Our study has set an a priori improvement of an absolute percentage change of 10% as significant. Using a single tail change in improvement (alpha = 0.025) with the intervention with an 80% power, we calculated the number needed for each cohort to be 291 subjects, however we will randomize for 360 in each cohort for a total of 720 subjects to allow for attrition.

Randomization:

Using the statistical package 'R', a series of random numbers will be generated to allocate individual patients to groups. This random number series will be validated for randomness using the 'runs test' available in SPSS. A conservative P value of 0.50 will be used to determine if the sequence of numbers is random. Randomization will continue until a sequence with a p-value greater than 0.50 is obtained. Once completed, the random number sequence will be saved to an Excel file and passed to Reading Hospital researchers for processing.

Data analysis:

Data analysis will occur in two separate phases. First descriptive analysis for all variables for patients within each group. For this analysis discrete variables will be reported as count, and percent within each category. For continuous variables statistics will include mean, minimum and maximum values, standard deviation and median. Significance testing will be conducted between groups. Discrete variables will use chi-square test and continuous variables will use group or independent t-test. An a priori p-value of 0.050 will determine statistical significance between groups.

The second phase of this analysis will include inferential statistics on the comparison between groups for both primary and secondary outcomes.

The primary outcomes to be compared between the PIVC insertion techniques include:

1. Failure rate (overall and individual cause/reason).
2. Utility time
3. Catheter-to-vein ratio

For the analysis of failure rate chi-square analysis will be used between the two groups. Utility time will be analyzed by group t-test. Catheter to vein ratio will be aggregated among all patients within group and a rate analysis defined by Fleiss will be used to determine if the ratios between treatment cohorts are significantly different. A standard p-value of 0.05 will be used for these analyses.

The secondary outcomes will be:

1. Describe post removal complication rates among traditional and US-guided PIVC insertion techniques
2. Identifying a catheter-to-vein ratio that predicts complication

The complication rate will be analyzed by standard rate analysis by Fleiss. Complication rates will be calculated as the number of complication divided by the number of patients.

In order to determine the catheter to vein ratio that may predict a complication, both groups will be added together in aggregate, and a ROC curve will be calculated using the catheter to vein ratio as the independent variable and the complication (0, 1) as the dependent variable. Standard methodology to determine the cutoff point will be used, (diagonal line drawn to ROC curve then projected down to sensitivity value) to determine the cutoff point. Standard ROC descriptive statistics will be used including area under the curve, standard error of the area, 95% confidence interval of the area, p-value as well as sensitivity and specificity of the cutoff value. The null hypothesis for the ROC curve will be area is equal to 0.50.

Due to the exploratory nature of these analysis there will be no corrections for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Identified as requiring a PIVC
* Acceptable vital signs - not requiring emergent resuscitation

Exclusion Criteria:

* Patients triaged as MI alert, brain attack alert, and trauma alert
* Pregnant
* Prisoners
* Institutionalized patients
* Housing insecurity
* Unable to provide consent
* Previously entered into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Post insertion failure rates | Duration of catheter dwell time (up to 168 hours)
  Failure rate (overall and individual cause/reason)
Overall utility | Up to 168 hours (1 week)
  The overall dwell time of the catheter

SECONDARY OUTCOMES:
Post removal complication rates | 48 hours after catheter removal
  Determining if ultrasound-guided peripheral intravenous catheter insertion results in lower post removal complication rates compared to PIVCs inserted in the standard manner.
Catheter to vein ratio | Up to 168 hours (1 week)
  Determining if catheter-to-vein ratio can predict post insertion success of PIVCs and what catheter-to-vein ratio is most successful. In this study, catheter-to-vein ratio is defined as the diameter of the lumen of the vein divided by the outside diameter of the catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Leroux, BS NRP, Principal Investigator — Reading Hospital
Locations (1):
- Reading Hospital, West Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braga LM, Parreira PM, Oliveira ASS, Monico LDSM, Arreguy-Sena C, Henriques MA. Phlebitis and infiltration: vascular trauma associated with the peripheral venous catheter. Rev Lat Am Enfermagem. 2018;26:e3002. doi: 10.1590/1518-8345.2377.3002. Epub 2018 May 17. PMID 29791668
- [Background] Helm RE, Klausner JD, Klemperer JD, Flint LM, Huang E. Accepted but unacceptable: peripheral IV catheter failure. J Infus Nurs. 2015 May-Jun;38(3):189-203. doi: 10.1097/NAN.0000000000000100. PMID 25871866
- [Background] Marsh N, Webster J, Larson E, Cooke M, Mihala G, Rickard CM. Observational Study of Peripheral Intravenous Catheter Outcomes in Adult Hospitalized Patients: A Multivariable Analysis of Peripheral Intravenous Catheter Failure. J Hosp Med. 2018 Feb 1;13(2):83-89. doi: 10.12788/jhm.2867. Epub 2017 Oct 18. PMID 29073316
- [Background] Murayama R, Uchida M, Oe M, Takahashi T, Oya M, Komiyama C, Sanada H. Removal of Peripheral Intravenous Catheters Due to Catheter Failures Among Adult Patients. J Infus Nurs. 2017 Jul/Aug;40(4):224-231. doi: 10.1097/NAN.0000000000000168. PMID 28683001
- [Background] Miliani K, Taravella R, Thillard D, Chauvin V, Martin E, Edouard S, Astagneau P; CATHEVAL Study Group. Peripheral Venous Catheter-Related Adverse Events: Evaluation from a Multicentre Epidemiological Study in France (the CATHEVAL Project). PLoS One. 2017 Jan 3;12(1):e0168637. doi: 10.1371/journal.pone.0168637. eCollection 2017. PMID 28045921
- [Background] Yabunaka K, Murayama R, Tanabe H, et al. Ultrasonographic classification of subcutaneous edema caused by infusion via peripheral intravenous catheter. Journal of Medical Ultrasound. 2016;24(2):60-5. doi: org/10.1016/j.jmu.2016.02.001
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Stolz LA, Stolz U, Howe C, Farrell IJ, Adhikari S. Ultrasound-guided peripheral venous access: a meta-analysis and systematic review. J Vasc Access. 2015 Jul-Aug;16(4):321-6. doi: 10.5301/jva.5000346. Epub 2015 Feb 4. PMID 25656255
- [Background] Tanabe H, Takahashi T, Murayama R, Yabunaka K, Oe M, Matsui Y, Arai R, Uchida M, Komiyama C, Sanada H. Using Ultrasonography for Vessel Diameter Assessment to Prevent Infiltration. J Infus Nurs. 2016 Mar-Apr;39(2):105-11. doi: 10.1097/NAN.0000000000000159. PMID 26934164
- [Background] Spencer TR, Mahoney KJ. Reducing catheter-related thrombosis using a risk reduction tool centered on catheter to vessel ratio. J Thromb Thrombolysis. 2017 Nov;44(4):427-434. doi: 10.1007/s11239-017-1569-y. PMID 29022210
- [Background] Nifong TP, McDevitt TJ. The effect of catheter to vein ratio on blood flow rates in a simulated model of peripherally inserted central venous catheters. Chest. 2011 Jul;140(1):48-53. doi: 10.1378/chest.10-2637. Epub 2011 Feb 24. PMID 21349931
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736